CLINICAL TRIAL: NCT05719038
Title: Construction of a Diagnostic and Prognostic Model of Pulmonary Fibrosis in Patients After COVID-19 Pneumonia and Study on Its Mechanism
Brief Title: Diagnostic and Prognostic Model of Pulmonary Fibrosis After COVID-19 Pneumonia and Mechanism Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuqi Cheng, Principal Investigator, Kunming Medical University
Other Study IDs: KunmingMC
Record Dates: First submitted 2023-02-05; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Fibrosis; COVID-19
MeSH Terms: conditions — Pulmonary Fibrosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group
  Interventions: Diagnostic Test: observational study
- Pulmonary fibrosis after COVID-19 Pneumonia
  Interventions: Diagnostic Test: observational study
- No pulmonary fibrosis after COVID-19 Pneumonia
  Interventions: Diagnostic Test: observational study

INTERVENTIONS:
Diagnostic Test: observational study — observational study

SUMMARY:
The infection of COVID-19 has caused serious threat to the life and health of all mankind and increased huge economic burden. According to the current statistics, the incidence of pulmonary fibrosis after COVID-19 infection is about 27.7% -87%, 81% of severe patients and 37% of moderate patients have residual lung lesions, and 53% of patients still have residual lung abnormalities one year after infection, resulting in restrictive pulmonary dysfunction and affecting the health and life of patients. Therefore, it is very important to study the diagnostic and prognostic markers of pulmonary fibrosis after infection of COVID-19. At present, relevant studies have been carried out on imagomics and serum proteomics of pulmonary fibrosis after COVID-19 infection, and serum biomarkers and imagomics marker models for diagnosing pulmonary fibrosis after COVID-19 pneumonia have been developed. However, there are few studies combining imageomics and serum proteomics, and the mechanism of pulmonary fibrosis after COVID-19 has not been fully clarified. In this study, it is planned to recruit patients with moderate, severe and critical COVID-19 pneumonia infection, collect venous blood from subjects, and perform chest HRCT follow-up. Blood samples were screened by proteomics and verified by expanded samples to screen diagnostic and prognostic markers of pulmonary fibrosis after COVID-19 infection. At the same time, based on deep learning technology, a model was developed to predict the occurrence and prognosis of pulmonary fibrosis after infection of COVID-19 combined with clinical characteristics, serum markers and AI imagomics, so as to provide ideas for further elucidating the mechanism of occurrence and development of pulmonary fibrosis after infection of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-90 years
2. novel coronavirus nucleic acid or antigen confirmed novel coronavirus infection
3. Meet the diagnostic criteria for moderate/severe/severe coronavirus infection in China (Trial Tenth Edition)
4. Chest CT showed that the extent of lung lesions was greater than 50%

Exclusion Criteria:

1. pregnant and lactating women
2. previous severe lung disease, such as known chronic lung disease: chronic obstructive pulmonary disease, asthma, interstitial lung disease, etc.
3. severe organ dysfunction: severe liver, kidney and heart dysfunction
4. severe epidemic defects (including tumors/severe rheumatism/organs, bone marrow transplantation/HIV, etc.)
5. inappropriate enrollment judged by the investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed COVID-19 pneumonia were classified as moderate, severe and critical according to clinical classification, and underwent chest CT imaging follow-up and blood protein measurement. In the later stage, patients were divided into groups with pulmonary fibrosis and without pulmonary fibrosis according to whether pulmonary fibrosis occurred; Healthy people as healthy control groups.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
change of pulmonary fibrosis | At the time of enrollment, The first month, the third month, the sixth month, the twelfth month
  The change of pulmonary fibrosis were evaluated

SECONDARY OUTCOMES:
change of protein in serum | At the time of enrollment, the third month
  Changes in plasma proteins over time
changes of Lung function | At the time of enrollment, the third month, the sixth month, the twelfth month
  Lung function over time

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xue M, Zhang T, Chen H, Zeng Y, Lin R, Zhen Y, Li N, Huang Z, Hu H, Zhou L, Wang H, Zhang XD, Sun B. Krebs Von den Lungen-6 as a predictive indicator for the risk of secondary pulmonary fibrosis and its reversibility in COVID-19 patients. Int J Biol Sci. 2021 Apr 10;17(6):1565-1573. doi: 10.7150/ijbs.58825. eCollection 2021. PMID 33907520
- [Result] Li X, Shen C, Wang L, Majumder S, Zhang D, Deen MJ, Li Y, Qing L, Zhang Y, Chen C, Zou R, Lan J, Huang L, Peng C, Zeng L, Liang Y, Cao M, Yang Y, Yang M, Tan G, Tang S, Liu L, Yuan J, Liu Y. Pulmonary fibrosis and its related factors in discharged patients with new corona virus pneumonia: a cohort study. Respir Res. 2021 Jul 9;22(1):203. doi: 10.1186/s12931-021-01798-6. PMID 34243776
- [Result] Yang J, Chen C, Chen W, Huang L, Fu Z, Ye K, Lv L, Nong Z, Zhou X, Lu W, Zhong M. Proteomics and metabonomics analyses of Covid-19 complications in patients with pulmonary fibrosis. Sci Rep. 2021 Jul 16;11(1):14601. doi: 10.1038/s41598-021-94256-8. PMID 34272434
- [Result] Sardar R, Sharma A, Gupta D. Machine Learning Assisted Prediction of Prognostic Biomarkers Associated With COVID-19, Using Clinical and Proteomics Data. Front Genet. 2021 May 20;12:636441. doi: 10.3389/fgene.2021.636441. eCollection 2021. PMID 34093642
- [Result] Bazdyrev E, Rusina P, Panova M, Novikov F, Grishagin I, Nebolsin V. Lung Fibrosis after COVID-19: Treatment Prospects. Pharmaceuticals (Basel). 2021 Aug 17;14(8):807. doi: 10.3390/ph14080807. PMID 34451904
- See also: Related Info — https://www.ijbs.com/v17p1565.htm
- See also: Related Info — https://respiratory-research.biomedcentral.com/articles/10.1186/s12931-021-01798-6
- See also: Related Info — https://www.nature.com/articles/s41598-021-94256-8
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fgene.2021.636441/full